CLINICAL TRIAL: NCT02890160
Title: A Randomized Trial of the Firesorb Sirolimus Target Eluting Bioresorbable Vascular Scaffold in Patients With Coronary Artery Disease: FUTURE-II
Brief Title: A Trial of Firesorb in Patients With Coronary Artery Disease: FUTURE-II
Acronym: FUTURE-II
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai MicroPort Medical (Group) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MicroPort_Firesorb_RCT
Record Dates: First submitted 2016-08-31; First posted 2016-09-07 (Estimated); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Coronary Artery Disease
Keywords: Bioresorbable Vascular Scaffold
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Firesorb (Experimental): Implantation of the Sirolimus Target Eluting Bioresorbable Vascular Scaffold （Firesorb）
  Interventions: Device: Firesorb
- XIENCE (Active Comparator): Implantation of the XIENCE Everolimus Eluting Coronary Stent System
  Interventions: Device: XIENCE

INTERVENTIONS:
Device: Firesorb — Sirolimus Target Eluting Bioresorbable Vascular Scaffold
  Arms: Firesorb
Device: XIENCE — Everolimus Eluting Coronary Stent System
  Arms: XIENCE

SUMMARY:
The FUTURE-II study is a confirmative clinical trial for Sirolimus Target Eluting Bioresorbable Vascular Scaffold (Firesorb) after the feasibility and safety of the device has been preliminary confirmed in a small-scale First-in-Man clinical trial.

DETAILED DESCRIPTION:
This study is a prospective, multicenter, single-blind, randomized controlled trial in patients with coronary artery disease caused by up to two de novo native coronary artery lesions in separate epicardial vessels. The goal is to evaluate the safety and effectiveness of Firesorb to support the approval of the Chinese Food and Drug Administration (CFDA) for this product. The Abbott's XIENCE Everolimus-eluting Coronary Stent System is selected as the control device. 430 subjects will be recruited. All subjects will be 1:1 randomly assigned to experimental group and control group. All subjects will undergo clinical follow-up at 1-month, 6-month, 1-year, 2-year, 3-year, 4-year and 5-year post-index procedure. All subjects will undergo angiographic follow-up at 1-year post-index procedure; of which 3-5 centers will be specified as a subgroup to complete OCT follow-up (n=80, 40 each in test and control group).

ELIGIBILITY:
General Inclusion Criteria:

1. 18-75 years of age, males or non-pregnant females;
2. With silent ischemia evidence, patients with stable or unstable angina, or in patients with old myocardial infarction;
3. Patients with indications for coronary artery bypass graft surgery;
4. To understand the purpose of testing, voluntary and informed consent, patients undergoing invasive imaging follow-up.

Angiographic Inclusion Criteria:

1. One or two de novo target lesions:

   1. If there is one target lesion, a second non-target lesion may be treated but the non-target lesion must be present in a different epicardial vessel, and must be treated first with a successful, uncomplicated result prior to randomization of the target lesion.
   2. If two target lesions are present, they must be present in different epicardial vessels and both must satisfy the angiographic eligibility criteria.
   3. The definition of epicardial vessels means the LAD, LCX and RCA and their branches. Thus, the patient must not have lesions requiring treatment in e.g. both the LAD and a diagonal branch.
2. Target lesion(s) must be located in a native coronary artery with a visually estimated or quantitatively assessed % diameter stenosis (DS) of ≥ 50% and < 100% with a thrombolysis in myocardial infarction (TIMI) flow of ≥1 and one of the following: stenosis ≥ 70%, an abnormal functional test (e.g. fractional flow reserve, stress test), unstable angina or post-infarct angina. Lesion(s) must be located in a native coronary artery with RVD by visual estimation of ≥ 2.5 mm and ≤4.0 mm. Lesion(s) must be located in a native coronary artery with length by visual estimation of ≤ 25 mm.
3. Each target lesion may be covered with one stent.

General Exclusion Criteria:

1. Within 1 week of any acute myocardial infarction or myocardial enzymes did not return to normal;
2. Implantation of stent in target vessel within 1 year , patients with planned intervention again within six months;
3. Severe congestive heart failure (NYHA III and above) ,or left ventricular ejection fraction <40% (ultrasound or left ventricular angiography);
4. Preoperative renal function serum creatinine >2.0mg/DL; receiving hemodialysis;
5. Bleeding, active gastrointestinal ulcers, brain hemorrhage or subarachnoid hemorrhage and half year history of ischemic stroke, antiplatelet agents and would not allow an anticoagulant therapy contraindications patients undergoing antithrombotic therapy;
6. Aspirin, clopidogrel, heparin, contrast agent, poly lactic acid polymer and rapamycin allergies;
7. The patient's life expectancy is less than 12 months;
8. Top participated in other drug or medical device and does not meet the primary study endpoint in clinical trials time frame;
9. Researchers determine patient compliance is poor, unable to complete the study in accordance with the requirements;
10. Heart transplantation patients;
11. The unstable arrhythmia, such as high risk ventricular extrasystole and ventricular tachycardia;
12. Cancer need chemotherapy;
13. Immunosuppression and autoimmune diseases, planned or undergoing immunosuppressive therapy;
14. Planning or being receiving long-term anticoagulant therapy, such as heparin, warfarin, etc;
15. Within six months for elective surgery requires stopping aspirin, Clopidogrel patients;
16. Blood test prompted platelet counts of less than 100x10E9/L or greater than 700x10E9/L, white blood cells than 3x10E9/L; known or suspected liver disease (such as hepatitis);
17. Peripheral vascular disease, 6F catheter is not available.

Angiographic Exclusion Criteria:

1. left main coronary artery disease;
2. severe triple vessel lesion and required revascularization.

The following exclusion criteria apply to the target lesion(s) or target vessel(s):

1. Aorto-ostial right coronary artery (RCA) lesion (within 3 mm of the ostium).
2. Lesion located within 3 mm of the origin of the Left Anterior Descending Artery (LAD) or left circumflex artery (LCX).
3. Lesion involving a bifurcation with a:

   1. side branch ≥ 2.5 mm in diameter, or
   2. side branch with diameter stenosis ≥ 50%, or
   3. side branch requiring guide wire, or
   4. side branch requiring dilatation.
4. Anatomy proximal to or within the lesion that may impair delivery of Firesorb or XIENCE stent:

   1. Extreme angulation (≥ 90°) proximal to or within the target lesion.
   2. Excessive tortuosity (≥ two 45° angles) proximal to or within the target lesion.
   3. Moderate or heavy calcification proximal to or within the target lesion.
5. Lesion or vessel involves a myocardial bridge.
6. Vessel contains thrombus as indicated in the angiographic images or by IVUS or OCT.
7. Vessel has been previously treated with a stent at any time prior to the index procedure such that the Firesorb or XIENCE would need to cross the stent to reach the target lesion.
8. Vessel has been previously treated and the target lesion is within 5 mm proximal or distal to a previously treated lesion.
9. Lesion which prevents successful balloon pre-dilatation, defined as full balloon expansion with the following outcomes:

   1. Residual %DS is a maximum of < 40% (per visual estimation), ≤ 20% is strongly recommended.
   2. TIMI Grade-3 flow (per visual estimation).
   3. No angiographic complications (e.g. distal embolization, side branch closure).
   4. No dissections National Heart Lung and Blood Institute (NHLBI) grade D-F.
   5. No chest pain lasting > 5 minutes.
   6. No ST depression or elevation lasting > 5 minutes.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Estimated)
Dates: Start 2017-08-24 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
In-segment Late Lumen Loss (LLL) (Queue 1) | 1 year after index procedure
  In-segment late lumen loss is defined as the change in minimal lumen diameter (MLD) within the margins of the scaffold/stent and 5mm proximal and 5mm distal to the scaffold/stent from post-procedure to 1 year by angiography.

SECONDARY OUTCOMES:
The percentage of intima coverage-strut (OCT subgroup) | 1 year after index procedure
  The main secondary endpoint
Vasomotion (Queue 2) | 2 year after index procedure
  The changes in average lumen diameter before and after intracoronary nitroglycerin
Acute Success-Device Success | From the start of index procedure to end of index procedure
  Successful delivery and deployment of the assigned scaffold/stent at the intended target lesion and successful withdrawal of the delivery system with attainment of final in-scaffold/stent residual stenosis of less than 30% by visual.
Acute Success-Procedural Success | At time of procedure up to 7 days in hospital
  Achievement of final in-scaffold/stent residual stenosis of less than 30% by visual estimation with successful delivery and deployment of at least one assigned scaffold/stent at the intended target lesion and successful withdrawal of the delivery system for the target lesion without the occurrence of cardiac death, target vessel MI or repeat TLR.
Device-oriented composite endpoints (Target Lesion Failure) | 1 month,6 months,1 year,2 years,3 years,4 years and 5 years after index procedure
  Target Lesion Failure is defined as the composited endpoints of cardiac death,target vessel myocardial infarction and clinical driven-target lesion revascularization.
Patient-oriented clinical composite endpoint (PoCE) | 1 month,6 months,1 year,2 years,3 years,4 years and 5 years after index procedure
  Patient-oriented clinical composite endpoint is defined as all cause death, all myocardial infarction, and any revascularization.
Death (Cardiac, Vascular, Non-cardiovascular) | 1 month,6 months,1 year,2 years,3 years,4 years and 5 years after index procedure
  Cardiac death (CD): Any death due to proximate cardiac cause (e.g. MI, low-output failure, fatal arrhythmia), unwitnessed death and death of unknown cause, all procedure related deaths including those related to concomitant treatment. Non-cardiovascular death: Any death not covered by the above definitions such as death caused by infection, malignancy, sepsis, pulmonary causes, accident, suicide or trauma.
Myocardial Infarction (MI) | 1 month,6 months,1 year,2 years,3 years,4 years and 5 years after index procedure
  Attributable to target vessel (TV-MI) Not attributable to target vessel (NTV-MI)
Target Vessel Revascularization (TVR) | 1 month,6 months,1 year,2 years,3 years,4 years and 5 years after index procedure
  Ischemia-driven TVR (ID-TVR) Not ischemia-driven TVR (NID-TVR)
Target Lesion Revascularization (TLR) | 1 month,6 months,1 year,2 years,3 years,4 years and 5 years after index procedure
  Ischemia-driven TLR (ID-TLR) Not ischemia-driven TLR (NID-TLR)
Any Revascularization | 1 month,6 months,1 year,2 years,3 years,4 years and 5 years after index procedure
Scaffold/Stent Thrombosis (per ARC definition) | 1 month,6 months,1 year,2 years,3 years,4 years and 5 years after index procedure
  Timing (acute, sub-acute, late and very late) Evidence (Definite and Probable)
Site Diagnosed Angina (SDA) | 1 month,6 months,1 year,2 years,3 years,4 years and 5 years after index procedure
  Defined as the study unit by collecting Seattle angina questionnaire (SAQ), doctor angina questionnaire and research units of AE reports incidence of angina pectoris (excludes angina pectoris 0-7 days after index procedure ).
Minimum Lumen Diameter (MLD) | 1 year and 2 years after index procedure
  Including in-scaffold/stent, in-segment lesion, the proximal 5mm of stent, and the distal 5mm of stent.
percentage of diameter stenosis (%DS) | 1 year and 2 years after index procedure
  Including in-scaffold/stent, in-segment lesion, the proximal 5mm of stent, and the distal 5mm of stent.
Angiographic Binary Restenosis (ABR) | 1 year and 2 years after index procedure
  Including in-scaffold/stent, in-segment lesion, the proximal 5mm of stent, and the distal 5mm of stent.
Late Lumen Loss (LLL) | 1 year and 2 years after index procedure
  Including in-scaffold/stent, in-segment lesion, the proximal 5mm of stent, and the distal 5mm of stent.
Acute Stent Recoil | Immediately after index procedure
Descriptive analysis of morphometric, lesion composition and scaffold strut data obtained with OCT | 1 year and 2 years after index procedure
  OCT endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Runlin Gao, MD, Principal Investigator — Fu Wai Hospital & National Center for Cardiovascular Diseases in China
Locations (1):
- Fu Wai Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jiang J, Li C, Chen D, Song L, Cui Z, Li P, Gan L, Chen Y, Li H, Jia S, He S, Lu W, Gao R, Wang J; FUTURE III Investigators. Firesorb bioresorbable scaffold for de novo coronary artery disease: 1-year clinical outcomes. BMC Med. 2025 Jul 9;23(1):419. doi: 10.1186/s12916-025-04254-0. PMID 40629329
- [Derived] Song L, Xu B, Chen Y, Zhou Y, Jia S, Zhong Z, Su X, Ma Y, Zhang Q, Liu J, Wang Y, Guan C, Zheng M, Qiao S, Gao R; FUTURE-II Trial Investigators. Thinner Strut Sirolimus-Eluting BRS Versus EES in Patients With Coronary Artery Disease: FUTURE-II Trial. JACC Cardiovasc Interv. 2021 Jul 12;14(13):1450-1462. doi: 10.1016/j.jcin.2021.04.048. Epub 2021 May 18. PMID 34238555